CLINICAL TRIAL: NCT07316348
Title: The Effcct of Vocalization and Spontaneous Pushing Techniqucs Used in Thc Second Stagc of Labour on Birth Outcomcs: A Randomised Controlled Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Yasemin Dincel, Researcher Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 26.2025fbu
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Second Stage of Labor; Maternal Pushing Techniques; Perineal Trauma; Maternal Fatigue
Keywords: Labor; Pain; Satisfaction; Perineal Trauma; Pushing
MeSH Terms: conditions — Pain; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM 2 (No Intervention): No specific instructions will be given regarding how the mother should push during the second stage of labor.
- ARM 1 (Experimental): During the second stage of labor, vocalization pushing techniques (using the vowels A, O, and U to exhale in deep tones) will be encouraged, and the mother's pushing will be observed.
  Interventions: Procedure: The vocalization straining technique will be used.

INTERVENTIONS:
Procedure: The vocalization straining technique will be used. — During the second stage of labor, vocalization pushing techniques (using the vowels A, O, and U to exhale in deep tones) will be encouraged, and the mother's pushing will be observed.
  Arms: ARM 1

SUMMARY:
The second stage of labor, defined as the period from full cervical dilatation to fetal birth, is a critical phase in which maternal pushing techniques may significantly affect maternal and neonatal outcomes (1-5). Evidence indicates that directed Valsalva pushing may be associated with maternal apnea, increased fatigue, pelvic floor injury, and adverse fetal effects, whereas spontaneous pushing with an open glottis supports physiological birth processes (2,5-11). The World Health Organization recommends encouraging women to follow their natural pushing urges and supports the use of open-glottis pushing techniques to promote a positive childbirth experience (12).

Vocalization pushing is an open-glottis maneuver involving intentional low-tone sound production during exhalation, which may facilitate pelvic floor relaxation, improve pain management, and enhance the birth experience (9-11). However, evidence regarding the effectiveness of vocalization pushing is limited, and data from Türkiye are lacking. This randomized controlled clinical trial aims to evaluate the effects of vocalization and spontaneous pushing techniques during the second stage of labor on labor duration, pain intensity, perineal trauma, maternal fatigue, and childbirth experience.

DETAILED DESCRIPTION:
The second stage of labor begins with complete cervical dilatation and continues until the birth of the fetus. During this phase, important physiological events occur, including increased contraction frequency and intensity, fetal descent, and rotation through the birth canal (2,5). Pushing is a physiological response that facilitates fetal expulsion through coordinated uterine contractions and maternal effort (2,5).

Two primary pushing techniques are described in the literature: Valsalva pushing, characterized by breath-holding with a closed glottis, and spontaneous pushing, performed with an open glottis following the woman's natural urge (2,3,5-9). Studies report that Valsalva pushing may lead to maternal apnea, increased fatigue, fetal head compression, pelvic floor damage, and impaired bladder function (2,7,10,11). In contrast, open-glottis pushing techniques have been associated with reduced maternal and fetal distress, protective effects on the perineum, decreased labor pain, shorter second-stage duration, higher Apgar scores, improved umbilical cord pH values, and greater maternal satisfaction (5,6,10-14).

Vocalization pushing, defined as intentional low-tone sound production (e.g., "A," "O," or "U") during exhalation, is a maneuver aimed at maintaining an open glottis during pushing (10,11). Evidence suggests that vocalization during childbirth may promote pelvic floor relaxation, reduce the severity of perineal lacerations, improve pain coping through vibrational effects, and contribute to a more positive and empowering birth experience (9-12). Despite these potential benefits, the literature contains limited high-quality evidence regarding vocalization pushing, and no clinical studies have examined its use during the second stage of labor in Türkiye.

This randomized controlled trial will compare vocalization pushing and spontaneous pushing techniques during the second stage of labor. Eligible women will be randomly assigned to either the vocalization pushing group or the spontaneous pushing group. Outcomes will include duration of the second stage of labor, pain intensity, perineal trauma, maternal fatigue, and childbirth experience. The findings are expected to support evidence-based, physiological, and woman-centered intrapartum care practices.

ELIGIBILITY:
Inclusion Criteria for the Study:

* Being 18 years of age or older
* Being nulliparous
* Being at term (between 38 and 42 weeks of gestation)
* Expecting a vaginal delivery
* Having a singleton pregnancy
* Presenting in vertex position
* Estimated fetal weight between 2500-4000 g
* Having had a complication-free pregnancy in terms of both mother and fetus
* Not having any perinatal risks
* Not having received any analgesia or anesthesia to relieve pain and fatigue during labor
* Being able to read, understand, and write Turkish
* Voluntarily agreeing to participate in the study

Exclusion Criteria:

* Being multiparous
* Having a multiple pregnancy
* Having dysphonia and hearing loss
* Being a high-risk pregnant woman
* Having any systemic, chronic, or neurological disease
* Pregnant women with fetal risk (presentation anomaly, cephalopelvic disproportion, macrosomia, SGA, fetal death, fetus without gross pathology according to ultrasound)

Endpoints for Cases Included in the Study:

* Loss of the baby during labor or delivery
* Delivery by cesarean section
* Pharmacological intervention to relieve pain and fatigue during labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 112 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Visuel Analog Scale -Pain | When cervical dilation is 8-9 cm and within the first 30 minutes after delivery
  Min: 0- Max:10
Birth Experience Scale | When cervical dilation is 8-9 cm and within the first 30 minutes after delivery
  Min: 42- Max:150
Visual Analogue Scale for Fatigue | When cervical dilation is 8-9 cm and within the first 30 minutes after delivery
  Min: 0- Max:10

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Dinçel, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University Cerrahpaşa, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sen E, Gunaydin S, Yilmaz T, Dinc Kaya H. The Effect of Music on Labor Pain and Duration: A Systematic Review and Meta-Analysis. Adv Mind Body Med. 2023 Fall;37(4):4-11. PMID 38466048
- [Result] Yilmaz T, Tas O, Gunaydin S, Kaya HD. The effect of Pilates on pain during pregnancy and labor: a systematic review and meta-analysis. Rev Assoc Med Bras (1992). 2023 Sep 18;69(10):e20230441. doi: 10.1590/1806-9282.20230441. eCollection 2023. PMID 37729226
- [Result] Dunmez F, Yilmaz T. The effect of using birth ball and squatting position during labor on pain, duration, and satisfaction: A randomized controlled trial. Jpn J Nurs Sci. 2024 Apr;21(2):e12580. doi: 10.1111/jjns.12580. Epub 2023 Dec 10. PMID 38073180
- [Result] Gunaydin S, Sen E, Yilmaz T, Kaya HD. Use of Transcutaneous Electrical Nerve Stimulation (TENS) in Labor Pain: An Integrative Review. Pain Manag Nurs. 2025 Feb;26(1):85-92. doi: 10.1016/j.pmn.2024.10.004. Epub 2024 Nov 12. PMID 39537497